CLINICAL TRIAL: NCT00455780
Title: Weight Loss Maintenance in Primary Care
Acronym: PrimaryCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Michael R. Lowe, Ph.D., Drexel University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DK66759 (completed); R01DK066759 (NIH)
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Obesity; Overweight
Keywords: Eating; Dieting; Meal replacements; Energy Density; Weight Loss Maintenance
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MR-/REDE- (Experimental): Weight Loss through cognitive behavioral therapy and meal replacement use, and continued therapy for weight loss maintenance.
  Interventions: Behavioral: Weight Loss Phase; Behavioral: Continued CBT
- MR+/REDE- (Experimental): Weight Loss through cognitive behavioral therapy and meal replacement use, and continued therapy and use of meal replacements for weight loss maintenance.
  Interventions: Behavioral: Weight Loss Phase; Behavioral: Continued CBT; Behavioral: continued use of meal replacements
- MR-/REDE+ (Experimental): Weight Loss through cognitive behavioral therapy and meal replacement use, and continued therapy as well as Reduced Energy Density Education for weight loss maintenance.
  Interventions: Behavioral: Weight Loss Phase; Behavioral: Continued CBT; Behavioral: reduced energy density education
- MR+/REDE+ (Experimental): Weight Loss through cognitive behavioral therapy and meal replacement use, and continued therapy, as well as Reduced Energy Density Education and continued meal replacement use, for weight loss maintenance.
  Interventions: Behavioral: Weight Loss Phase; Behavioral: Continued CBT; Behavioral: reduced energy density education; Behavioral: continued use of meal replacements

INTERVENTIONS:
Behavioral: Weight Loss Phase — Weight loss using CBT and meal replacements
Behavioral: Continued CBT — Using CBT during weight loss maintenance
Behavioral: reduced energy density education — Additional nutritional learning
  Arms: MR+/REDE+; MR-/REDE+
Behavioral: continued use of meal replacements — continued use of meal replacements during weight loss maintenance
  Arms: MR+/REDE+; MR+/REDE-

SUMMARY:
After a three month weight loss phase involving the use of meal replacements, participants are randomized into different weight loss maintenance conditions. Aim 1: To test the hypothesis that the meal replacement (MR) and reduced energy density eating (REDE) interventions, when added separately to the LEARN program, will produce superior weight loss maintenance compared to a LEARN-only intervention. Aim 2: To test the hypothesis that the weight loss maintenance condition that combines MRs and REDE will produce better maintenance of weight losses than either individual component and than the LEARN-only condition. Aim 3: To test the hypothesis that the two conditions receiving the REDE intervention will experience longer-lasting improvements in the energy density and nutritional composition of the diet compared to the two non-REDE conditions.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 30, or BMI of 27 with weight-related comorbidities
* Access to a telephone and voice mail/answering machine
* MUST be seeing a primary care physician working with us on this study (in the greater Philadelphia area)

Exclusion Criteria:

* Previously/currently diagnosed with an eating disorder
* Current bi-polar, depression, substance abuse, or dependence disorder
* Living with someone already enrolled
* Enrolled in another weight loss program
* Current disorder/medications affecting body weight or energy expenditure (e.g. thyroid disease)
* Myocardial infraction within the past three months
* Unstable angina
* Nephrotic syndrome/malabsorptive disease
* Gout attack within the past year
* Lactating/pregnant (or planning within next two years)
* Current/recent history of cancer, neurological disease, high creatinine levels, active hepatic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2005-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Weight | baseline, 3 months, 12 months, 24 months, 36 months

SECONDARY OUTCOMES:
Body composition | baseline, 3 months, 12 months, 24 months, 36 months
Blood work results | baseline, 3 months, 12 months, 24 months
Scores on questionnaire-based measures | baseline, 3 months, 12 months, 24 months, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Lowe, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States